CLINICAL TRIAL: NCT03206788
Title: Losartan as Anti-inflammatory Therapy to Augment F508del Cystic Fibrosis Transmembrane (CFTR) Recovery
Brief Title: Losartan and Inflammation in Cystic Fibrosis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: due to slow enrollment and approval of the Trikafta for CF patients
Sponsor: University of Miami (Other)
Collaborators: University of Alabama at Birmingham (Other); Children's Hospital Medical Center, Cincinnati (Other); University of Kansas Medical Center (Other); Cystic Fibrosis Foundation (Other)
Responsible Party: Principal Investigator, Matthias Salathe, Emeritus Professor, University of Miami
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20170397; 20170333 (Other: Human Subject Research Office at University of Miami)
Record Dates: First submitted 2017-06-29; First posted 2017-07-02 (Actual); Results first posted 2020-11-13 (Actual); Last update posted 2020-11-27 (Actual); Status verified 2020-11

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — Losartan

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Losartan group (Experimental): Participant will receive the Losartan intervention and will take 50 mg losartan orally once daily for week 1, followed by 50 mg orally twice daily on weeks 2-12 (unless weight adjustment needed).
  Interventions: Drug: Losartan
- Placebo group (Placebo Comparator): Participant will receive the placebo intervention, matching the Losartan intervention, once daily for week 1, followed by twice daily on weeks 2-12.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Losartan — 25 mg or 50 mg (based on patient's weight) Losartan tablets taken by mouth daily in the morning for week 1 followed by twice daily (one in the morning and one in the evening) on Weeks 2-12.
  Other Names: Cozaar
  Arms: Losartan group
Drug: placebo — Placebo tablets, matching the Losartan intervention, taken by mouth daily in the morning for week 1 followed by twice daily (one in the morning and one in the evening) on Weeks 2-12.
  Other Names: matching placebo twice daily
  Arms: Placebo group

SUMMARY:
The purpose of the study is to examine if a specific drug called losartan (Cozaar ®), generally used to treat high blood pressure and to protect kidneys from damage in patients suffering from Diabetes Mellitus, will have any effect on the nasal inflammation in patients with cystic fibrosis (CF). The study will be performed at the Pulmonary Division at the University of Miami, Cincinnati Children's Medical Hospital Center, University of Kansas Medical Center and University of Alabama-Birmingham.

ELIGIBILITY:
Inclusion Criteria:

* CF patients homozygous for F508del and on current treatment with Orkambi™ for at least 3 months
* Age >12 years
* Forced expiratory volume at one second (FEV1) >/= 40% of predicted

Exclusion Criteria:

* Female patients not willing to adhere to strict birth control (combination of two methods)
* Pregnancy
* History of intolerance to angiotensin receptor blockers (ARBs)
* Treatment with angiotensin converting enzyme (ACE) inhibitor
* NPD response to zero chloride (0Cl)/isoproterenol of > - 6.6 mV at screening (evidence of detectable CFTR activity at baseline)
* Regular use of NSAIDs or potassium supplementation, treatment with aliskiren, on anticoagulation
* Oral corticosteroid use within 6 weeks
* Exacerbation requiring treatment within 6 weeks
* Active treatment for mycobacterial infections
* Significant hypoxemia (oxygen saturation <90% on room air and rest or use of continuous oxygen treatment), chronic respiratory failure by history (pCO2 > 45 mmHg), clinical evidence of cor pulmonale
* Untreated arterial hypertension (systolic blood pressure >140 mm Hg, diastolic blood pressure > 90 mmHg)
* Blood pressure less than 90 mm Hg systolic while standing
* Cardiac, renal (creatinine 1.5 times normal limit), hepatic (LFTs > 3x normal upper limit), neurological, psychiatric, endocrine or neoplastic diseases that are judged to interfere with participation in study
* Known renal artery stenosis
* Concomitant airway disorders other than CF, such as allergic bronchopulmonary aspergillosis (ABPA).
* Subjects with prior thoracic surgery

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2017-11-11 (Actual); Primary Completion 2019-10-24 (Actual); Study Completion 2019-12-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Salathe, MD, Principal Investigator — University of Miami
Locations (4):
- United States (4):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of Miami, Miller School of Medicine, Miami, Florida
  - University of Kansas, Kansas City, Kansas
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Losartan Group | Placebo Group
Started | 2 | 5
Completed | 2 | 2
Not Completed | 0 | 3
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Adverse Event | 0 | 1
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Losartan Group | Placebo Group | Total
Number analyzed (Participants) | 2 | 5 | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 5 | 7
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 | 2
  Male | 2 | 3 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 2 | 4 | 6
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 2 | 5 | 7
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Nasal Potential Difference (NPD) to Assess CFTR Activity
Description: Cystic Fibrosis Transmembrane Conductance Regulator (CFTR) activity will be measured as the change in NPD in response to apical perfusion with 0 Cl-/isoproterenol. NPD will be measured at the nasal epithelium via a voltmeter.
Time Frame: Baseline, 12 weeks
Measure: Mean (Standard Error); unit: mV
Arm/Group | Losartan Group | Placebo Group
Number analyzed (Participants) | 2 | 2
mV | -4.2 (2.1) | 1.59 (2.48)

2. Secondary Outcome: Change in NPD to Assess CaCC Activity
Description: Potential difference of Calcium dependent Chloride Channels (CaCC) will be measured as the change in NPD on on Adenosine Triphosphate (ATP) stimulation. NPD will be measured at the nasal epithelium via a voltmeter.
Time Frame: Baseline, 12 weeks
Measure: Mean (Standard Error); unit: mV
Arm/Group | Losartan Group | Placebo Group
Number analyzed (Participants) | 2 | 2
mV | 2.14 (1) | -5.43 (7.1)

3. Secondary Outcome: Change in NPD to Assess BK Activity
Description: Big Potassium (BK) activity will be measured as the change in NPD on Adenosine Triphosphate (ATP) stimulation. NPD will be assessed from nasal epithelium samples and analyzed via a voltmeter.
Time Frame: Baseline, 12 weeks
Measure: Mean (Standard Error); unit: mV
Arm/Group | Losartan Group | Placebo Group
Number analyzed (Participants) | 2 | 2
mV | 2.14 (1) | -5.43 (7.1)

4. Secondary Outcome: Change in FEV1
Description: Forced Expiratory Volume in 1 second (FEV1) assessed in liters will be measured using spirometry.
Time Frame: Baseline, 12 weeks
Measure: Mean (Standard Error); unit: Liter
Arm/Group | Losartan Group | Placebo Group
Number analyzed (Participants) | 2 | 2
Liter | -0.18 (0.18) | 1.85 (0.1)

5. Secondary Outcome: Change in Sweat Chloride Concentration
Description: Sweat chloride concentration will be analyzed from participant sweat samples analyzed in millimoles per liter (mmol/l)
Time Frame: Baseline, 12 weeks
Measure: Mean (Standard Error); unit: mmol/l
Arm/Group | Losartan Group | Placebo Group
Number analyzed (Participants) | 2 | 2
mmol/l | -2.5 (7.5) | -3 (6)

6. Secondary Outcome: Change in Quality of Life (QoL) Scores as Assessed by the CFQ-R
Description: Cystic Fibrosis Questionnaire-Revised (CFQ-R) is a quality of life questionnaire with a total score ranging from 0-100 with a higher score indicating increased quality of life.
Time Frame: Baseline, 12 weeks
Population: Values were not measured for this outcome for all participants.
Arm/Group | Losartan Group | Placebo Group
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Change in Cytokine Levels
Description: Nasal airway epithelial cells taken by brush will be assessed for cytokine levels including Interleukin IL-1beta, Transforming Growth Factor (TGF-beta) active and total, IL-6, IL-8 and IL-13 in pg/mL.
Time Frame: Baseline, 12 weeks
Population: Values were not measured for this outcome for all participants.
Arm/Group | Losartan Group | Placebo Group
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Change in hsCRP
Description: Serum samples will be analyzed for High sensitivity C-Reactive Protein (hsCRP) values in mg/L.
Time Frame: Baseline, 12 weeks
Population: Values were not measured for this outcome for all participants.
Arm/Group | Losartan Group | Placebo Group
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Change in Blood Count Values
Description: Serum blood count values including white blood count (WBC) and Absolute Neutrophil Counts (ANC) will be evaluated in units/uL.
Time Frame: Baseline, 12 weeks
Population: Values were not measured for this outcome for all participants.
Arm/Group | Losartan Group | Placebo Group
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Change in %PMN Values
Description: Serum samples will be analyzed for % Polymorphonuclear (PMN) cells.
Time Frame: Baseline, 12 weeks
Population: Values were not measured for this outcome for all participants.
Arm/Group | Losartan Group | Placebo Group
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Change in SAA Values
Description: Serum samples will be analyzed for Serum Amyloid A (SAA) values in mg/L.
Time Frame: Baseline, 12 weeks
Population: Values were not measured for this outcome for all participants.
Arm/Group | Losartan Group | Placebo Group
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Change in Calprotectin Values
Description: Serum samples will be analyzed for calprotectin values in ug/mg.
Time Frame: Baseline, 12 weeks
Population: Values were not measured for this outcome for all participants.
Arm/Group | Losartan Group | Placebo Group
Number analyzed (Participants) | 0 | 0

13. Secondary Outcome: Change in GM-CSF Values
Description: Serum samples will be analyzed for % Granulocyte/Macrophage Colony Stimulating Factor (GM-CSF) values in pg/mL.
Time Frame: Baseline, 12 weeks
Population: Values were not measured for this outcome for all participants.
Arm/Group | Losartan Group | Placebo Group
Number analyzed (Participants) | 0 | 0

14. Secondary Outcome: Change in TGF-beta Values
Description: Serum samples will be analyzed for TGF-beta values in ng/mL.
Time Frame: Baseline, 12 weeks
Population: Values were not measured for this outcome for all participants.
Arm/Group | Losartan Group | Placebo Group
Number analyzed (Participants) | 0 | 0

15. Secondary Outcome: Change in mRNA Expression
Description: Change in messenger ribonucleic acid (mRNA) expression from nasal cells evaluated via quantitative polymerase chain reaction (qPCR) for Leucine Rich Repeating Protein 26 (LRRC26) and TGF-Beta).
Time Frame: Baseline, 12 weeks
Population: Values were not measured for this outcome for all participants.
Arm/Group | Losartan Group | Placebo Group
Number analyzed (Participants) | 0 | 0

16. Secondary Outcome: Change in Losartan Metabolites Levels
Description: Change in serum blood levels of Losartan and Losartan metabolites EXP3179 & EXP3174.
Time Frame: Baseline, 12 weeks
Population: Values were not measured for this outcome for all participants.
Arm/Group | Losartan Group | Placebo Group
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 16 weeks
Arm/Group | Losartan Group | Placebo Group
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/5
Other Adverse Events (participants affected / at risk) | 2/2 | 5/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Losartan Group (N=2) | Placebo Group (N=5)
nose bleed (General disorders) | 1 (2) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
muscle cramps (Musculoskeletal and connective tissue disorders) | 1 (2) | 1 (5)
Sore throat (General disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 3 (5)
Fatigue (General disorders) | 0 (0) | 1 (1)
Pulmonary exacerbation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-02-01): https://cdn.clinicaltrials.gov/large-docs/88/NCT03206788/Prot_SAP_000.pdf